CLINICAL TRIAL: NCT00968019
Title: A Multicenter Postmarket Surveillance Registry Evaluating the Performance and Long Term Safety of the Presillion Stent in de Novo Native Coronary Artery Lesions. Iberian Registry
Brief Title: Multicenter Postmarket Surveillance Registry Evaluating Performance and Long Term Safety of the Presillion Stent
Status: Completed | Type: Observational
Sponsor: Johnson and Johnson, S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: 08-CR-001
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Results first posted 2013-03-06 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Coronary Arteriosclerosis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Presillion stent: Patients treated with the Presillion stent in up to two de novo coronary artery lesions
  Interventions: Device: Presillion stent

INTERVENTIONS:
Device: Presillion stent — Centers will use commercially available Presillion Stents as recommended according to the Instruction For Use (IFU).

SUMMARY:
The purpose of this study is: To evaluate the safety and performance of the Presillion stent in routine clinical practice.

DETAILED DESCRIPTION:
Primary endpoint: Composite of Major Adverse Cardiac Events (MACE), which includes cardiac death, myocardial infarction (Q-wave and non Q-wave) and clinically driven target lesion revascularization (TLR) at 12 months follow-up.

Data will be collected on 400 patients (from 14 hospitals in Spain and Portugal) treated with the Presillion stent in up to 2 de novo native coronary artery lesions

Study design: multicenter, prospective, observational

ELIGIBILITY:
Inclusion Criteria:

* All subjects treated with Presillion stent up to two de novo coronary artery lesions

Exclusion Criteria:

* No specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All sujects treated with Presillion stent up to two de novo coronary artery lesions
Sampling Method: Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2009-04; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angel Cequier, MD, PhD, Principal Investigator — Hospital Universitario de Bellvitge
Locations (13):
- Portugal (4):
  - Hospital Garcia Da Orta, Almada
  - Hospital de Santa Cruz, Lisbon
  - Hospital Sao Joao, Porto
  - Centro Hospitalar Vila Real, Vila Real
- Spain (9):
  - Complejo Hospitalario Universitario de Albacete, Albacete, Albacete
  - Hospital Germans Trias I Pujol, Badalona, Barcelona
  - Centro Medico Teknon, Barcelona, Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Capio Hospital General de Cataluña, Sant Cugat del Vallès, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Arnau de Vilanova, Lleida, Lerida
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias

RESULTS

PARTICIPANT FLOW:
Groups:
- Treated With Presillion Stent: Patients treated with the Presillion stent in up to two de novo coronary artery lesions
Period: Overall Study
Arm/Group | Treated With Presillion Stent
Started | 318
Completed | 303
Not Completed | 15

BASELINE CHARACTERISTICS:
Arm/Group | Treated With Presillion Stent
Number analyzed (Participants) | 318
Age Continuous [Mean (Standard Deviation); unit: years] | 65.5 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 248
Region of Enrollment [Number; unit: participants]
  Portugal | 56
  Spain | 262

OUTCOME MEASURES:

1. Primary Outcome: Major Cardiac Adverse Events (Including Cardiac Death, Myocardial Infarction (Q-wave and Non Q-wave) and Clinically Driven TLR (Target Lesion Revascularization))
Description: Major adverse cardiac and cerebral events are defined as an adjudicated composite of cardiac death, myocardial infarction (Q-wave and non Q-wave), emergent coronary artery bypass surgery and target vessel revascularization (TVR).
  The primary safety measure was the composite of MACE up to 12 months follow up. In order to show the safety of the device, the MACE rate was compared with the performance goal for bare metal stents(experience with bare metal stents in clinical trials suggested that the 12 month MACE rate should be about 25.0%).
Time Frame: at 12 months follow-up
Population: No formal statistical significance testing was performed. Descriptive statistics were calculated for all relevant variables (mean, standard deviation, median and ranges for the continuous variables and with frequencies and % for the discrete variables). Subjects who discontinued prematurely were included in the analysis and were not replaced.
Measure: Number; unit: participants
Arm/Group | Treated With Presillion Stent
Number analyzed (Participants) | 308
participants | 9

2. Secondary Outcome: Device Success
Description: Device success defined as achievement of a final diameter stenosis of <50% (by visual estimate), using the assigned device only
Time Frame: Peri-procedure up to discharge
Population: 318 patients treated with the Presillion stent in up to two de novo coronary artery lesions (354 lesions)
Measure: Number; unit: percentage of device success
Units Other Than Participants: Lesions
Arm/Group | Treated With Presillion Stent
Number analyzed (Participants) | 318
Number analyzed (Lesions) | 354
percentage of device success | 98.9

3. Secondary Outcome: Lesion Success
Description: Lesion success defined as the attainment of <50% final diameter stenosis (by visual estimate) using any percutaneous method.
Time Frame: Peri-procedure up to discharge
Population: 318 patients treated with the Presillion stent in up to two de novo coronary artery lesions (354 lesions)
Measure: Number; unit: percentage of lesion Success
Units Other Than Participants: Lesion
Arm/Group | Treated With Presillion Stent
Number analyzed (Participants) | 318
Number analyzed (Lesion) | 354
percentage of lesion Success | 98.6

4. Secondary Outcome: Procedural Success
Description: Procedural success defined as achievement of a final diameter stenosis of <50% (by visual estimate) using any percutaneous method, without the occurrence of death, MI (Myocardial Infarction), or repeat revascularization of the target lesion during the hospital stay
Time Frame: Peri-procedure up to discharge
Population: 318 patients treated with the Presillion stent in up to two de novo coronary artery lesions (354 lesions)
Measure: Number; unit: percentage of Procedural Success
Units Other Than Participants: Lesions
Arm/Group | Treated With Presillion Stent
Number analyzed (Participants) | 318
Number analyzed (Lesions) | 354
percentage of Procedural Success | 97.2

5. Secondary Outcome: Clinically Driven TLR
Description: Target Lesion Revascularization (TLR) is defined as any clinically-driven repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel
Time Frame: Up to 30 days
Population: 309 patients treated with the Presillion stent in up to two de novo coronary artery lesions (311 lesions)
Measure: Number; unit: participants
Units Other Than Participants: Lesions
Arm/Group | Treated With Presillion Stent
Number analyzed (Participants) | 309
Number analyzed (Lesions) | 311
participants | 2

6. Secondary Outcome: Clinically Driven TVR
Description: Target vessel revascularization (TVR) is defined as any clinically driven (as defined for TLR) repeat percutaneous intervention of the target vessel or bypass surgery of the target vessel.
Time Frame: Up to 30 days
Population: 309 patients treated with the Presillion stent in up to two de novo coronary artery lesions (311 lesions)
Measure: Number; unit: participants
Units Other Than Participants: Lesions
Arm/Group | Treated With Presillion Stent
Number analyzed (Participants) | 309
Number analyzed (Lesions) | 311
participants | 2

7. Secondary Outcome: Target Vessel Failure
Description: Target vessel failure includes any target vessel revascularization as well as any MI or any cardiac death that cannot be clearly attributed to a non-target vessel.
  Target vessel failure will be reported when:
  1. MI occurs in territory not clearly attributed to a vessel other than the target vessel.
  2. Cardiac death not clearly due to a non-target vessel endpoint.
  3. Target vessel revascularization is performed.
Time Frame: Up to 30 days
Population: 309 patients treated with the Presillion stent in up to two de novo coronary artery lesions (311 lesions)
Measure: Number; unit: participants
Units Other Than Participants: Lesions
Arm/Group | Treated With Presillion Stent
Number analyzed (Participants) | 309
Number analyzed (Lesions) | 311
participants | 7

8. Secondary Outcome: Myocardial Infarction
Description: A positive diagnosis of myocardial infarction is made when one of the following criteria is met:
  1. Typical rise and/or fall of biochemical markers of myocardial necrosis together with evidence of ischemia with at least one of the following:
     * ischemic symptoms
     * ECG changes indicative of ischemia (ST segment elevation or depression)
     * Development of pathological Q waves in the ECG
     * Imaging evidence of new an equivocal loss of viable myocardium or new regional wall motion abnormality
  2. Pathological findings of an acute myocardial infarction
Time Frame: Up to 30 days
Population: 309 patients treated with the Presillion stent in up to two de novo coronary artery lesions (311 lesions)
Measure: Number; unit: participants
Units Other Than Participants: Lesions
Arm/Group | Treated With Presillion Stent
Number analyzed (Participants) | 309
Number analyzed (Lesions) | 311
participants | 6

9. Secondary Outcome: Major Bleeding
Time Frame: Up to 30 days
Measure: Number; unit: participants
Arm/Group | Treated With Presillion Stent
Number analyzed (Participants) | 309
participants | 0

10. Secondary Outcome: Stroke
Time Frame: Up to 30 days
Measure: Number; unit: participants
Arm/Group | Treated With Presillion Stent
Number analyzed (Participants) | 309
participants | 0

11. Secondary Outcome: Stent Thrombosis
Description: Thrombosis is defined as the formation of blood clot derived from aggregation of red cells or platelets obstructing the lumen of the vessel.
Time Frame: Up to 30 days
Measure: Number; unit: participants
Arm/Group | Treated With Presillion Stent
Number analyzed (Participants) | 309
participants | 2

12. Secondary Outcome: Clinically Driven TLR
Description: as for outcome 5
Time Frame: up to 12 months
Population: 303 patients treated with the Presillion stent in up to two de novo coronary artery lesions (308 lesions)
Measure: Number; unit: participants
Units Other Than Participants: Lesions
Arm/Group | Treated With Presillion Stent
Number analyzed (Participants) | 303
Number analyzed (Lesions) | 308
participants | 5

13. Secondary Outcome: Clinically Driven TVR
Description: as for outcome 6
Time Frame: Up to 12 months
Population: 303 patients treated with the Presillion stent in up to two de novo coronary artery lesions (308 lesions)
Measure: Number; unit: participants
Units Other Than Participants: Lesions
Arm/Group | Treated With Presillion Stent
Number analyzed (Participants) | 303
Number analyzed (Lesions) | 308
participants | 5

14. Secondary Outcome: Target Vessel Failure
Description: as for outcome 7
Time Frame: Up to 12 months
Population: 303 patients treated with the Presillion stent in up to two de novo coronary artery lesions (308 lesions)
Measure: Number; unit: participants
Units Other Than Participants: Lesions
Arm/Group | Treated With Presillion Stent
Number analyzed (Participants) | 303
Number analyzed (Lesions) | 308
participants | 11

15. Secondary Outcome: Myocardial Infarction
Description: as for outcome 8
Time Frame: Up to 12 months
Population: 303 patients treated with the Presillion stent in up to two de novo coronary artery lesions (308 lesions)
Measure: Number; unit: participants
Units Other Than Participants: Lesions
Arm/Group | Treated With Presillion Stent
Number analyzed (Participants) | 303
Number analyzed (Lesions) | 308
participants | 8

16. Secondary Outcome: Major Bleeding
Time Frame: Up to 12 months
Measure: Number; unit: participants
Arm/Group | Treated With Presillion Stent
Number analyzed (Participants) | 303
participants | 0

17. Secondary Outcome: Stent Thrombosis
Description: as for outcome 11
Time Frame: Up to 12 months
Measure: Number; unit: participants
Arm/Group | Treated With Presillion Stent
Number analyzed (Participants) | 303
participants | 2

18. Secondary Outcome: Stroke
Time Frame: Up to 12 months
Measure: Number; unit: participants
Arm/Group | Treated With Presillion Stent
Number analyzed (Participants) | 303
participants | 0

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | Treated With Presillion Stent
Serious Adverse Events (participants affected / at risk) | 39/318
Other Adverse Events (participants affected / at risk) | 17/318
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated With Presillion Stent (N=318)
Mortality (General disorders) | 5 (5)
Myocardial infarction (Cardiac disorders) | 8 (8)
Revascularization (Vascular disorders) | 13 (13)
Bleeding or vascular event (Vascular disorders) | 4 (4)
Serious Adverse Events not related to the study device (General disorders) | 9 (9)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated With Presillion Stent (N=318)
Signs that do not interfere, or interferes but does not hinder, with the subject's usual activity (General disorders) | 17 (17)

LIMITATIONS AND CAVEATS:
since the difference with the performance goal is this large; the possibility of underreporting of adverse events is something that needs to be considered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No